CLINICAL TRIAL: NCT04265079
Title: I2-CoRT WTP9 Bovenste Extremiteit Motoriek Interventie Met Hand Orthese Bij Mensen na Een Beroerte
Brief Title: I2-CoRT WTP9: Upper Extremity Motor Intervention, Use of Hand Orthosis in People Post-stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study could not be executed due to COVID-19 regulations.
Sponsor: Maastricht University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I2-CoRT_WTP9_BEMIHOMB
Record Dates: First submitted 2020-01-22; First posted 2020-02-11 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Upper Extremity Dysfunction
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Masking Description: Study focusses on within participant comparison and cannot be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Added weight to hand (Experimental)
  Interventions: Other: Additional weight at hand

INTERVENTIONS:
Other: Additional weight at hand — Added weight of an inactive hand orthosis (300 gram)

SUMMARY:
The upper extremity kinematics of people post-stroke will be monitored with/without an inactive hand orthosis (intervention: added weight to hand) during ARAT, Fugl-Meyer, and Box and Blocks tests. Measurements will occur right after inclusion and repeated once after 7-8 weeks. Upper extremity kinematics and test scores will indicate the influence of additional weight to hand as a possible confounder when, in the future, the hand orthosis would be used as a therapy tool.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke
* Receive regular therapy at Jessa hospital
* Able to willingly sign informed consent

Exclusion Criteria:

* Relapse during study
* Secundary complications limiting upper extremity performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test | 0 weeks
  Score
Action Research Arm Test | 8 weeks
  Score
Fugl-Meyer | 0 weeks
  Score
Fugl-Meyer | 8 weeks
  Score
Box and Blocks | 0 weeks
  Score
Box and Blocks | 8 weeks
  Score
Upper extremity kinematics | 0 weeks
  Joint angles
Upper extremity kinematics | 8 weeks
  Joint angles

IPD SHARING:
Plan to Share IPD: Undecided